CLINICAL TRIAL: NCT05000723
Title: Long Term Follow-up of Patients With Prosthetic Joint Infection of the Hip Treated at University Hospitals Leuven
Acronym: PROFITH
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S65804
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Prosthetic Joint Infection; Hip Prosthesis Infection
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PJI patients: Patients (older than 18 years) with PJI of a total hip replacement treated at University Hospitals Leuven.
  Diagnosis of PJI of the hip is made based on the EBJIS 2021 criteria. Patients will receive standard of care.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Standard of care consisting of
  * clearance of infection
  * treatment with antibiotics (antisuppressive, DAIR) or surgery (1 stage, 2 stage Girdlestone)
  * Radiology: X-ray pelvis and hip, X-ray pelvis with kingmark, CT scan pelvis/hip

SUMMARY:
Prosthetic Joint Infection (PJI) of a Total Hip Replacement (THR) is a disastrous complication of an otherwise extremely successful surgical procedure. It is associated with a burdensome treatment for the patient, significant challenges for the medical team and high costs for society. As more joint replacements are being performed each year, due to an ageing population and lower thresholds for surgery, the number of PJIs is on the rise. Many of these patients will be referred to University Hospitals Leuven as the physicians have extensive experience with this particular pathology and can offer a multidisciplinary and patient-tailored treatment. Many controversies exist in the field of PJI treatment, both with regard to the surgical aspects as well as the antibiotic treatment. Setting up randomized controlled trials to answer these questions has been proven to be very difficult due to large variations in patients, implants, germs, soft and hard tissues, antibiotic resistance patterns, and so on. Also, surgery for PJIs is usually non-elective / semi-urgent and therefore time to include patients into different trials is limited. Therefore the investigators will prospectively collect data on patients with PJI treated at University Hospitals Leuven, starting 01/01/2022, in order to have knowledge of own results and inform patients about chances of success prior to treatment; perform internal audits and quality checks; answer questions in the field of PJI treatment not suitable for RCTs.

DETAILED DESCRIPTION:
Prosthetic Joint Infection (PJI) of a Total Hip Replacement (THR) is a disastrous complication of an otherwise extremely successful surgical procedure. It is associated with a burdensome treatment for the patient, significant challenges for the medical team and high costs for society. As more joint replacements are being performed each year, due to an ageing population and lower thresholds for surgery, the number of PJIs is on the rise. Many of these patients will be referred to University Hospitals Leuven as the physicians have extensive experience with this particular pathology and can offer a multidisciplinary and patient-tailored treatment.

Many controversies exist in the field of PJI treatment, both with regard to the surgical aspects as well as the antibiotic treatment. Setting up randomized controlled trials to answer these questions has been proven to be very difficult due to large variations in patients, implants, germs, soft and hard tissues, antibiotic resistance patterns, and so on. Also, surgery for PJIs is usually non-elective / semi-urgent and therefore time to include patients into different trials is limited.

Nevertheless, prospectively collecting data on patients with PJI who are not involved in RCTs can already be helpful. It would allow the investigators to provide the patients with percentages of success of certain interventions based on historical results. At the moment the investigators have to rely on results reported by other groups, who might use different techniques or a facing a different germ spectrum.

Furthermore, prospectively collecting data on this cohort of patients, would make it possible for the investigators to do internal audits for quality control. Being able to perform simple checks, for example is every patient discussed in the multi-disciplinary team meeting, or is the hospital switching to targeted antibiotics soon enough, would already add to the quality of the service and could lead to adjustments in the protocols.

Also, certain scientific questions, which do not lend themselves to RCTs, such as the rate of success of treatment of PJI caused by rare germs (e.g. fungi) or in a specific population (e.g. octogenarians, transplant patients), could be answered by maintaining a prospective database

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* patients diagnosed with PJI of the hip based on EBJIS 2021 criteria

Exclusion Criteria:

* Patients unable to provide written informed consent
* Patients who prefer treatment outside of University Hospitals Leuven
* Patients with infections of the native hip joint
* Patients with fracture-related infections (FRI)
* Patients with uncertain diagnosis of PJI according to the 2021 EBJIS criteria
* Patient younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every adult patient (> 18 years), regardless of sex or age, with a PJI of the hip, as based on the EBJIS 2021 criteria, is eligible for inclusion on this study. This would therefore also include women of childbearing age, although this would be extremely rare.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2099-12 (Estimated); Study Completion 2099-12 (Estimated)

PRIMARY OUTCOMES:
Clearance of infection | within 5 years
  Clearance of infection based on DELPHI criteria

SECONDARY OUTCOMES:
Chosen treatment strategy | within 5 years
  description of chosen treatments strategy such as suppressive antibiotics, Debridement Antibiotics Implant Retention (DAIR), 1 stage, 2 stage, Girdlestone
Surgical complications | within 5 years
  Occurence of sugical complications such as fracture, dislocation, nerve damage, bleeding
Medical complications | within 5 years
  Occurence of complications such as delirium, renal failure, deep venous thrombosis, hospital acquired pneumonia
Length of hospital stay | within 5 years
  length of hospital stay in days
Discussion of patient in multi-disciplinary meeting | within 5 years
  Whether or not patient is discussed in multi-disciplinary meeting
Readmissions within 30 days | within 30 days
  Occurence of readmissions within 30 days
Mortality | within 5 years
  Mortality of patients
EuroQol 5D -3L | within 5 years
  Patients Reported Outcome Measures
General treatment discussion | within 5 years
  Appropriate work-up performed? Unnecessary aspirations? Unnecessary nuclear imaging?
Hip disability and Osteoarthritis Outcome Score | within 5 years
  Patients Reported Outcome Measures
Western Ontario and McMaster Universities Osteoarthritis Index | within 5 years
  Patients Reported Outcome Measures
Readmissions within 90 days | within 90 days
  Occurence of readmissions within 90 days
Changes in treatment | within 5 years
  Whether or not there are changes in treatment consequent to multi-disciplinary meeting

CONTACTS AND LOCATIONS:
Overall Officials: Georges Vles, Md, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven - Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No